CLINICAL TRIAL: NCT01379079
Title: Aspirin AM or PM in Reduction of Tension: a Randomized Cross-over Trial
Brief Title: Aspirin in Reduction of Tension II Study
Acronym: ASPIRETENSION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Principal Investigator, J.G. vd Bom, MD, PhD, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL34954.058.10; 2010-024448-13 (EudraCT Number); P10.246 (Other: Leiden University Medical Center)
Record Dates: First submitted 2011-03-31; First posted 2011-06-23 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Aspirin; carbaspirin calcium; acetylsalicylic acid lysinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aspirin at bedtime (Experimental)
  Interventions: Drug: Acetylsalicylic acid
- aspirin on awakening (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid lysinate

INTERVENTIONS:
Drug: Acetylsalicylic acid — aspirin intake at bedtime
  Other Names: Ascal, Ascal Cardio/Neuro, Carbasalate Calcium
  Arms: aspirin at bedtime
Drug: Acetylsalicylic acid lysinate — aspirin intake on awakening
  Other Names: Ascal, Ascal Cardio/Neuro, Carbasalate Calcium
  Arms: aspirin on awakening

SUMMARY:
Aspirin is a cornerstone in the secondary prevention of cardiovascular disease (CVD) and is usually taken on awakening, although evidence regarding optimal time of intake is lacking. Recent studies in healthy subjects with mild hypertension showed that aspirin at bedtime decreases blood pressure (-7/5mmHg), whereas intake of aspirin on awakening does not. Additionally, the investigators found that aspirin at bedtime decreases plasma renin activity, catecholamines and cortisol over 24hrs. Time-dependent effects of aspirin have never been studied in patients with CVD, who may use concomitant antihypertensive drugs. Moreover, platelet reactivity has a circadian rhythm, and intake of aspirin at bedtime may attenuate the morning peak in platelet reactivity. The investigators hypothesize that aspirin intake at bedtime compared with on awakening decreases both blood pressure and platelet reactivity over 24h.

A randomized open-label blinded endpoint crossover trial in which 250 patients, recruited from primary care, will be included who use aspirin for secondary prevention of CVD and have a stable blood pressure of 149/94mmHg or lower. Study subjects will randomly use both aspirin on awakening and at bedtime during two intervention periods of three months. Blood pressure will be recorded for 24hrs at the end of each treatment period in the patients' normal daily situation. To assess effects on platelet inhibition, thromboxane-B2 levels will be measured in a 24h urine sample at the end of both treatment periods. The investigators will asses differential effects according to time of intake on gastrointestinal complaints and potential minor bleeding events, as well as compliance.

The aim of this study is to evaluate the effect of aspirin taken at bedtime compared with on awakening on blood pressure of subjects with stable CVD. In addition, it will generate insights into the effect of aspirin on platelet reactivity over 24hrs, potential side effects and compliance.

DETAILED DESCRIPTION:
Aspirin is a cornerstone in the secondary prevention of cardiovascular disease because of its inhibitory effects on platelet aggregation. It reduces the risk of recurrent cardiovascular events with about a quarter. Although not supported by evidence, aspirin is usually taken at morning. There are several reasons why it may be more beneficial to take aspirin at bedtime instead of on awakening. First, one of the most important modifiable risk factors for cardiovascular disease is arterial hypertension. Aspirin is usually assumed to have no effects on blood pressure. However, in two randomized clinical trials of Hermida et al. among (otherwise healthy) grade I hypertensive subjects (140/90-159/99 mmHg), aspirin intake at bedtime decreased 24h blood pressure with 6.8/4.6 and 7.2/4.9 mmHg, whereas use of aspirin at morning slightly increased blood pressure (2.6/1.6 and 1.3/0.8 mmHg). The investigators have demonstrated that aspirin at bedtime decreases both plasma renin activity over 24h and excretion of catecholamines and cortisol in 24h urine compared to morning intake. Decreased activity of these pressor systems forms a biologically plausible explanation for the finding that aspirin at bedtime may reduce blood pressure whereas aspirin at morning does not. The effect of aspirin at bedtime versus on awakening on blood pressure has never been studied in a clinically relevant group of patients, i.e. patients already using aspirin for the secondary prevention of recurrent atherothrombotic events who mostly use also a wide variety of concomitant (antihypertensive) drugs. If time of intake has an effect, this could lead to a very simple improvement of therapy at no extra cost. Second, it has been convincingly shown that there is a morning peak in platelet reactivity, which might partly explain the increase in cardiovascular events in the early morning (highest incidence between 6 and 12 AM). Coming in an upright posture can lead to increased platelet activity and platelets can also be stimulated by the early morning increase of sympathetic activity (which starts few hours before awakening). Since platelet reactivity has a circadian rhythm, time of intake of aspirin may influence its inhibitory effect on platelets. It has been argued that intake of aspirin at bedtime could better prevent the early morning increase in platelet reactivity than intake at morning assuming that intake at morning would be too late.

The aim of our project is to study whether treatment with aspirin at bedtime compared with intake at morning has additional benefits in patients using aspirin to prevent recurrent cardiovascular events. Our primary objective is to study the effect of 100 mg aspirin intake at bedtime compared with 100 mg aspirin intake at morning on blood pressure (24h ambulatory blood pressure measurements (ABPM)) in patients who use aspirin for secondary prevention of recurrent atherothrombotic events. As a secondary objective, the investigators will study the effect of aspirin intake at bedtime compared with at morning on platelet function. Furthermore, the investigators will address differential effects on potential side effects and compliance, as well as potential effect modification of the effect on blood pressure by genes involved in blood pressure regulation.

ELIGIBILITY:
Inclusion Criteria:

* Use of low-dose aspirin (acetylsalicylic acid or carbasalate calcium 80- 100mg [brand names: acetylsalicylic acid cardio, aspirin protect, ascal cardio, carbasalate calcium cardio]) for secondary prevention of cardiovascular events
* Stable blood pressure (with or without therapy) between 120/70 and 159/99
* Age 18-80 year
* Capacity to give informed consent (IC)

Exclusion Criteria:

* Blood pressure lower than 120/70 or higher than 159/99
* Change in blood pressure lowering medication within the last three months
* Regular use of non-steroidal anti-inflammatory drugs (NSAID's)
* Shift workers
* Evidence of secondary arterial hypertension
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
change in 24h Ambulant blood pressure measurement | after 3 and 6 months
  Primary endpoint: 24-hour Ambulatory blood pressure (ABPM). The primary endpoint will be analysed in primary- and secondary analysis. Primary analysis population: all randomized subjects with complete follow-up ABPM. Includes subjects with invalid ABPM, change in antihypertensive medication during follow-up, and subjects with low compliance. Analyses: 1) paired t-tests: mean 24-hour blood pressure, blood pressure during the day and night. 2)Linear mixed models: timing of aspirin intake, treatment sequence, treatment period, used blood pressure device and interaction terms as fixed effects, and subjects as random effects. Secondary analysis population excludes subjects with invalid ABPM, change of antihypertensive medication, or compliance <90%. Subgroup analyses: 1) β-blockers: yes/no; 2)Ace-inhibitors: yes/no; 3)Subjects using: a.No β-blockers or Ace-inhibitors; b.β-blockers; c. Ace-inhibitors; d. β-blockers+Ace-inhibitors; 4)Office blood pressure <140/90 mmHg vs. >140/90 mmHg.

SECONDARY OUTCOMES:
Platelet inhibition | after 3 and 6 months
  Secondary endpoint: Platelet reactivity measured during morning hours in a subsample (n=160). Primary analysis: paired t-test to compare means in platelet reactivity after the interventions. Additionally, a relative decrease/increase in platelet reactivity, to facilitate comparison with other studies in this field and evaluate clinical relevance. Subgroup analyses:we defined the following subgroups for analysis: 1)Diabetics vs non-diabetics; 2)Smokers vs non smokers; 3)High mean platelet volume (MPV) vs. low MPV.
platelet function and coagulation factors | baseline and after 3 and 6 months
  Platelet function and factors involved in coagulation- and fibrinolytic pathways, measured in blood samples.
side effects | baseline and after 3 and 6 months
  side effects of aspirin intake on awakening or at bedtime
genes involved in blood pressure regulation | baseline
Patient preference | baseline and after 6 months
  Baseline use of aspirin and preference of timing of Aspirin use after completion of the study was assessed by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: J.G. vd Bom, MD, PhD, Study Director — Leiden University Medical Center; T.N. Bonten, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Snoep JD, Hovens MM, Pasha SM, Frolich M, Pijl H, Tamsma JT, Huisman MV. Time-dependent effects of low-dose aspirin on plasma renin activity, aldosterone, cortisol, and catecholamines. Hypertension. 2009 Nov;54(5):1136-42. doi: 10.1161/HYPERTENSIONAHA.109.134825. Epub 2009 Oct 5. PMID 19805643
- [Background] Hermida RC, Ayala DE, Calvo C, Lopez JE. Aspirin administered at bedtime, but not on awakening, has an effect on ambulatory blood pressure in hypertensive patients. J Am Coll Cardiol. 2005 Sep 20;46(6):975-83. doi: 10.1016/j.jacc.2004.08.071. PMID 16168278